CLINICAL TRIAL: NCT07042633
Title: Mechanism of Gamma Oscillation Synchronization in the Prefrontal-hippocampal Circuit for Memory Dysfunction in Patients With White Matter Lesions of Cerebral Small Vessel Disease
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: NO.2024092
Record Dates: First submitted 2025-05-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Vascular Cognitive Impairment; White Matter Lesions; Gamma Oscillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The mechanism underlying memory impairment caused by white matter lesions of cerebral small vessel disease is still unclear. The disrupted synchronization of gamma oscillations in the prefrontal-hippocampal circuit is a potential key mechanism. Our study has demonstrated that white matter lesions lead to demyelination of the connection tracts between the prefrontal lobe and hippocampus, which is closely related to memory dysfunction. However, further studies are required to explore if these microstructural changes in white matter tracts influence memory function by affecting gamma oscillations. Thus, this project will use the previously established episodic memory task and event-related potential to determine the changes in gamma oscillations in the prefrontal-hippocampal circuit and the effects on memory encoding and retrieval. Combining multimodal imaging, we will explore the mediating role of white matter microstructure damage, and establish a machine learning prediction model for memory impairment. In addition, transcranial alternation current stimulation (tACS) will be used to investigate the mechanisms of memory improvement by regulating the prefrontal-hippocampal gamma oscillations. This project will clarify the neural oscillation mechanism underlying memory impairment caused by white matter lesions of cerebral small vessel disease, with the expectation of providing new predictive indicators and interventions.

ELIGIBILITY:
Inclusion Criteria:

* - Individuals with cerebral small vessel disease, normal cognition or mild cognitive impairment subjects;
* Participants with complete demographic data, neuropsychiatric scale assessments, imaging data, and EEG data.

Exclusion Criteria:

* Severe aphasia, physical disability, or other conditions preventing completion of neuropsychological assessments;
* History of cerebrovascular stroke with documented neurological deficits during onset and corresponding lesions on neuroimaging;
* Neurological disorders that may cause cognitive impairment, including alcohol abuse, drug addiction, traumatic brain injury, epilepsy, encephalitis, or normal-pressure hydrocephalus;
* Systemic diseases potentially contributing to mild cognitive impairment (e.g., hepatic/renal insufficiency, endocrine disorders, vitamin deficiencies);
* Current diagnosis of major depressive disorder or psychiatric disorders.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly population
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall cognitive function | baseline and one-year follow-up
  Mini-Mental State Examination (MMSE) and the Montreal Cognitive Assessment (MOCA) scale scores.

SECONDARY OUTCOMES:
Attention and executive functions | Baseline and follow up
  the scores are evaluated using the Clock Drawing Test (CDT), the Digit Span Test (DST), and the Trail Making Test (TMT).
Language function | Baseline and one-year follow up
  Boston Naming Test (BNT)
Memory function | Baseline and one-year follow up
  Digit Span Test (DST) and the WHO-UCLA Auditory Verbal Learning Test (AVLT).
Brain imaging data | baseline and one-year follow-up
  Based on DTI data, the following metrics can be extracted:
  Fractional Anisotropy (FA) Mean Diffusivity (MD) Axial Diffusivity (AD) Radial Diffusivity (RD)
Electroencephalogram (EEG) data. | baseline and one-year follow-up
  Based on EEG data, time-frequency analysis and cross-frequency coupling analysis can be performed to extract the following metrics:
  Theta Band Neural Oscillation Energy Theta-Gamma Coupling Strength

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China